CLINICAL TRIAL: NCT05015543
Title: Glioblastoma and Sports - Does a Personal Training Program Improve Physical Performance and Quality of Life of Brain Tumor Patients
Brief Title: Physical Training in Glioblastoma Patients During Cytotoxic Therapy
Acronym: MMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MMH_01
Record Dates: First submitted 2021-06-23; First posted 2021-08-20 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Glioblastoma
Keywords: sports; Glioblastoma (GBM); physical training; Quality of Life (QOL); Neuro-Oncology; Psycho-Oncology; fitness
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients paticipating in the Personal Training Program (Experimental): The study patients complete two training sessions per week (60 minutes each) under supervision (16 weeks)
  Interventions: Other: Personal Training Program

INTERVENTIONS:
Other: Personal Training Program — One training sessions includes an interval training on a bicycle ergometer. The second one is a strength training with exercise machines. Both trainings are supplemented by coordinative aspects.

SUMMARY:
The aim of the present study is the prospective controlled use of physical activity in a collective of patients with glioblastoma after surgery and concomitant radiation/chemotherapy and during adjuvant cytotoxic therapy. The research question is whether physical exercise is feasible and whether patients benefit physically and mentally from the activities performed. For this purpose, specific training units under the supervision of a certified trainer and sports scientist as well as standardized sports medical test procedures are implemented. Beyond the instructed training, general physical activity phases are recorded electronically using a pedometer/activity tracker, which is worn at all times.

It will be examined whether the individual training program

1. improves physical fitness
2. increases quality of life/life satisfaction throughout the intervention
3. can be detected in blood due to increased concentrations of brain-derived neurotrophic factor 1 (BDNF-1) (voluntary)

The measurements should be taken before and 8, 16 and 24 weeks after the start of training.

DETAILED DESCRIPTION:
The personal trainers of the university clinics in Bochum and Homburg/Saar receive specific training activities from Münster's trainer Ralf Brandt in order to ensure a standardized concept. This way, a comparison of the trainings' conduction and recording is possible both quantitatively and qualitatively.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed glioblastoma
* Karnofsky Index ≥ 70
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* ≥ 18 years
* Completed surgical therapy
* Completed radiation and chemotherapy
* Thrombocytes > 50.000/µl
* Hb > 8 mg/dl
* Ability to give consent
* Mother tongue German/very good German skills

Exclusion Criteria:

* Diagnosed dementia (Mini-Mental-State-Test < 24/30 points)
* Pain (strong, permanent, restricting movement)
* Impairment of consciousness
* Fever
* Acute infection
* Pregnancy and lactation
* Insufficiently adjusted epilepsy (despite anticonvulsive therapy > 3 focal seizures per day or > 1 generalized seizure in the previous 3 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Increase in Physical Performance according to Physical Work Capacity (PWC) Test | Between week 0 and 16.
  Evidence of a significant increase (at least 15%) in physical work [watt/kilogram bodyweight] at PWC75% of maximum heart rate.

SECONDARY OUTCOMES:
Physical Work Capacity (PWC) | Between week 0 and 16 (and 24).
  PWC stratified according to:
  * age (<40, 40-60, >60 years)
  * Karnofsky performance status (KPS) (70-80 vs. 90-100 %)
  * Gender
  * PWC test 130, 150, (170)
PWC | after 8, 16 and 24 weeks
  changes over time, follow-up
Spiroergometry - maximal oxygen consumption (VO2max) | Between week 0 and 16 (and 24).
  Changes in the maximal oxygen consumption (measured during spiroergometry)
Spiroergometry - lactate | Between week 0 and 16 (and 24).
  Changes in the individual anaerobic lactate threshold (measured during spiroergometry)
EORTC-QLQ-C30 Brain module | Between week 0 and 16 (and 24).
  Changes in Health Related Quality of Life (HRQoL) using a standardized questionnaire; The EORTC QLQ-C30 questionnaire contains 30 questions and assesses the quality of life of oncology patients multidimensionally across 10 subscales. Times of measurement in week 0, 4, 8, 16, 20 and 24.
Distress Thermometer (DT) | Between week 0 and 16 (and 24).
  Changes in Health Related Quality of Life (HRQoL) using a standardized questionnaire; scale from 1 (not stressed at all) to 10 (extremly stressed); Times of measurement in week 0, 4, 8, 16, 20 and 24.
Hospital Anxiety and Depression Scale (HADS) | Between week 0 and 16 (and 24).
  Changes in Health Related Quality of Life (HRQoL) using a standardized questionnaire; The Hospital Anxiety and Depression Scale (HADS) is a self-rating scale developed to assess psychological distress in non-psychiatric patients. It consists of two subscales, anxiety and depression (14 items); Times of measurement in week 0, 4, 8, 16, 20 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothee Wiewrodt, PD Dr. med., Principal Investigator — Universitätsklinikum Münster
Locations (1):
- Universitätsklinikum Münster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No